CLINICAL TRIAL: NCT06417905
Title: Effects Of Exercise Training On Core Endurance, Scapular And Upper Exstremity Functions in Dentists
Brief Title: Effect of Exercises on Dentists' Body Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Emrullah ALKAN, Msc, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: supervisedvsvideovscontrol
Record Dates: First submitted 2024-05-13; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Neck Pain
Keywords: muscle strength; muscle endurance; pain; neck pain; musculoskeletal problems
MeSH Terms: conditions — Neck Pain; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supervised Exercises (Experimental): Exercises were done 3 times a week for 12 weeks with a physiotherapist
  Interventions: Other: Supervised exercises
- Video based Exercises (Experimental): Exercises were done 3 times a week for 12 weeks by subjects via videos
  Interventions: Other: video based exercises
- Control Group (No Intervention): Only postural education were given

INTERVENTIONS:
Other: Supervised exercises — strengthening deep neck flexors, serratus anterior middle and lower trapez stretchening upper trapezius, levator scapula
  Arms: Supervised Exercises
Other: video based exercises — strengthening deep neck flexors, serratus anterior middle and lower trapez stretchening upper trapezius, levator scapula
  Arms: Video based Exercises

SUMMARY:
The aim of the study is to compare the effects of supervised exercises, video based exercises and control group on muscle strength, muscle endurance, pain and upper extremity function in dentists with musculoskeletal pain. Participants were randomly divided into 3 groups: Supervised exercise group (SEG), video based exercise group (VEG) and control group (CG). Both SEG and VEG were given same exercises but SEG did the exercises with a experienced physiotherapist while VEG did it through videos 3 days a week for 12 weeks. CG was only given postural education.

ELIGIBILITY:
Inclusion Criteria:

* working as an active dentist for at least 3 years
* Having nonspecific neck pain more than 3 months

Exclusion Criteria:

* any operation in neck area

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2024-01-25 (Actual)

PRIMARY OUTCOMES:
Change in pain | Before training and after 12 weeks of training
  change in pain was assessed by using algometer

SECONDARY OUTCOMES:
change in deep cervical flexor and extensor muscle endurance | Before training and after 12 weeks of training
  change in cervical flexor and extensor muscle endurance was assessed by physiotherapist
change in scapular muscle endurance | Before training and after 12 weeks of training
  change in scapular muscle endurance was assessed by physiotherapist
change in core static and dynamic endurance | Before training and after 12 weeks of training
  change in core static and dynamic endurance was assessed by physiotherapist
functional assessment | Before training and after 12 weeks of training
  functional assessment was assessed using DASH Questtionnaire
neck disability | Before training and after 12 weeks of training
  neck disability was assessed using neck disability index

CONTACTS AND LOCATIONS:
Locations (1):
- Dokuz Eylul University, Izmir, Turkey (Türkiye)